CLINICAL TRIAL: NCT05705518
Title: Effects Of Artificial Tears on Tear Lipid Films and Tear Film Dynamics In Vivo
Brief Title: Artificial Tears, Tear Lipids and Tear Film Dynamics
Acronym: AlconAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPHS_2022-09-15617
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye
Keywords: Dry Eye; Tear Film Lipid Layer Dynamics; Tear Film Stability
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: After the 1-week initial period during which all subjects will use the run-in solution, subjects will be randomly assigned one of the 4 study solutions, and neither the subject nor the clinician researchers or technicians conducting examinations and taking measurements will be aware of which solution is assigned. All 4 solutions will be dispensed in color- and name-coded identical dispensing bottles prepared by study personnel not involved in collecting data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Systane Complete PF (Treatment) (Experimental): Masked subjects assigned to Arm 1 will use Systane Complete PF artificial tear drops 4 times per day (QID) to treat dry eye symptoms over a 3 month period.
  Interventions: Drug: Systane Complete PF
- Refresh Relieva PF (Control) (Placebo Comparator): Masked subjects assigned to Arm 2 will use Refresh Relieva PF artificial tear drops 4 times per day (QID) to treat dry eye symptoms over a 3 month period.
  Interventions: Drug: Refresh Relieva PF
- Refresh Optive Mega-3 PF (Active Comparator 1) (Active Comparator): Masked subjects assigned to Arm 3 will use Refresh Optive Mega-3 PF artificial tear drops 4 times per day (QID) to treat dry eye symptoms over a 3 month period.
  Interventions: Drug: Refresh Optive Mega-3 PF
- CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2) (Active Comparator): Masked subjects assigned to Arm 4 will use CVS Health Lubricant Eye Drop (PG 0.6%) artificial tear drops 4 times per day (QID) to treat dry eye symptoms over a 3 month period.
  Interventions: Drug: CVS Health Lubricant Eye Drop (PG 0.6%)

INTERVENTIONS:
Drug: Systane Complete PF — 3 month use, 4 times daily, of Systane Complete PF, a lipid-based, preservative-free artificial tear product
  Arms: Systane Complete PF (Treatment)
Drug: Refresh Relieva PF — 3 month use, 4 times daily, of Refresh Relieva PF, a non-lipid-based, preservative-free artificial tear product
  Arms: Refresh Relieva PF (Control)
Drug: Refresh Optive Mega-3 PF — 3 month use, 4 times daily, of Refresh Optive Mega-3 PF, a lipid-based, preservative-free artificial tear product
  Arms: Refresh Optive Mega-3 PF (Active Comparator 1)
Drug: CVS Health Lubricant Eye Drop (PG 0.6%) — 3 month use, 4 times daily, of CVS Health Lubricant Eye Drop (PG 0.6%), a lipid-based, preserved artificial tear product
  Arms: CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2)

SUMMARY:
Dry eye disease (DED) is pervasive with some reports estimating over 16 million adults diagnosed in the United States. Currently, artificial tears remain an integral part of managing dry eyes and are mainly used for symptomatic relief. Recent studies have shown there may be therapeutic benefits with regular use of lipid-based artificial tears to improve the structure of the tear film, which may improve tear film stability and provide relief of symptoms. In this study the investigators propose to compare effects on the tear lipid film and its dynamics between 3 lipid based artificial tears and a widely available non-lipid based artificial tear.

DETAILED DESCRIPTION:
This is a prospective, double-masked, randomized, controlled, parallel-group trial designed to compare the impact of Systane Complete PF lipid-based artificial tears (the Treatment solution under study) on tear lipid layer thickness compared with a non-lipid Control solution, Refresh Relieva PF. Secondarily, the study will compare changes in tear lipid layer thickness, lipid layer uniformity, tear film thinning dynamics, and symptoms between the Treatment solution, the non-lipid Control solution, and 2 other available lipid-based solutions (Active Comparators: Refresh Optive Mega-3 PF and CVS Health Lubricant Eye Drop (PG 0.6%)). The study will include 4 clinic visits, and require 1 week of single-masked run-in with Systane Ultra PF (an over-the-counter non-lipid-based solution) followed by 3 months of study treatment dosing. All subjects will complete a screening interview, then an in-clinic baseline ocular health examination and study eligibility determination followed by dispensing of the Control solution to all subjects for 1 week of run-in. After that week, subjects will be randomized to 1 of the 4 artificial tear solutions and have an in-clinic ocular examination and dispense of the assigned solution to use for 3 months. An in-clinic follow-up examination is completed after 1 month of study solution use, followed by a phone interview at 2 months, and a final in-clinic examination at 3 months post-dispensing.

ELIGIBILITY:
Inclusion Criteria:

* Best Corrected Visual Acuity of 20/30 or better;
* Experiencing Dry Eye symptoms (baseline OSDI score >= 13);

Exclusion Criteria:

* Currently experiencing active ocular inflammation or infection;
* Currently using topical eye medication (not including over-the-counter eyedrops);
* Having systemic health conditions or using prescription medications (including but not limited to isotretinoin derivatives) that could alter tear film physiology;
* Having a history of severe ocular trauma, ocular surgery, or diabetes;
* Being pregnant or breast feeding;
* Being a current contact lens wearer;
* Currently having a condition or being in a situation which, in the examiner's opinion, may put the subject at significant risk, may confound the study results, or may otherwise significantly interfere with their participation in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng C. Lin, OD, PhD, Principal Investigator — University of California Berkeley Clinical Research Center
Locations (1):
- Clinical Research Center, School of Optometry, University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data collected in this study may be shared upon request, at the discretion of the PI, for non-commercial research purposes.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects participated in a 1-week run-in period during which they used a common over-the-counter non-lipid artificial tear (Systane Ultra PF). Upon completion of the run-in period, participants were then randomized to one of the 4 study solutions.
Groups:
- Run-in Period Participants: All subjects participate in a 1-week run-in period during which they used a common over-the-counter non-lipid artificial tear (Systane Ultra PF). Upon completion of the run-in period, participants will then be randomized to one of the 4 study solutions.
Period: 1-week Run-in Period
Arm/Group | Run-in Period Participants | Systane Complete PF (Treatment) | Refresh Relieva PF (Control) | Refresh Optive Mega-3 PF (Active Comparator 1) | CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2)
Started | 81 | 0 | 0 | 0 | 0
Completed | 81 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Post-run-in Period
Arm/Group | Run-in Period Participants | Systane Complete PF (Treatment) | Refresh Relieva PF (Control) | Refresh Optive Mega-3 PF (Active Comparator 1) | CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2)
Started | 0 | 18 | 21 | 19 | 23
Completed | 0 | 18 | 21 | 19 | 23
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Systane Complete PF (Treatment) | Refresh Relieva PF (Control) | Refresh Optive Mega-3 PF (Active Comparator 1) | CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2) | Total
Number analyzed (Participants) | 18 | 21 | 19 | 23 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (16.1) | 34.0 (16.6) | 38.4 (17.1) | 35.5 (17.3) | 36.0 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 16 | 16 | 59
  Male | 7 | 5 | 3 | 7 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity Group: Asian | 10 | 11 | 3 | 11 | 35
  Race/Ethnicity Group: Non-Asian | 8 | 10 | 16 | 12 | 46

OUTCOME MEASURES:

1. Primary Outcome: Tear Lipid Layer Thickness
Description: Change in Tear Lipid Layer Thickness (3mo follow-up - post-run-in baseline)
Time Frame: Lipid Layer Thickness measured once at post-run-in baseline and once at 3mo follow-up visit
Measure: Mean (95% Confidence Interval); unit: nm
Arm/Group | Systane Complete PF (Treatment) | Refresh Relieva PF (Control) | Refresh Optive Mega-3 PF (Active Comparator 1) | CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2)
Number analyzed (Participants) | 18 | 21 | 19 | 23
nm | 0.72 [-2.48 to 3.93] | -7.58 [-11.46 to -3.70] | 2.06 [-0.83 to 4.95] | 1.41 [-1.50 to 4.32]

2. Secondary Outcome: Tear Lipid Layer Uniformity
Description: Change (3mo follow-up - post-run-in baseline) in Tear Lipid Layer Thickness Coefficient of Variation (CV). The CV is calculated as the standard deviation divided by the mean lipid layer thickness. A greater value of the CV indicates more variability in lipid layer thickness, a smaller value of the CV indicates a more uniformly thick lipid layer.
Time Frame: Lipid Layer Uniformity measured once at post-run-in baseline and once at 3mo follow-up visit
Measure: Mean (95% Confidence Interval); unit: Unitless
Arm/Group | Systane Complete PF (Treatment) | Refresh Relieva PF (Control) | Refresh Optive Mega-3 PF (Active Comparator 1) | CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2)
Number analyzed (Participants) | 18 | 21 | 19 | 23
Unitless | -0.15 [-0.66 to 0.37] | -0.77 [-1.47 to -0.06] | -0.01 [-0.58 to 0.56] | -0.23 [-0.70 to 0.24]

3. Secondary Outcome: Tear Film Thinning Rate
Description: Change in Tear Film Thinning rate (3mo follow-up - post-run-in baseline)
Time Frame: Tear Film Thinning Rate measured once at post-run-in baseline and once at 3mo follow-up visit
Measure: Mean (95% Confidence Interval); unit: % Area of Fluorescein Darkening / sec
Arm/Group | Systane Complete PF (Treatment) | Refresh Relieva PF (Control) | Refresh Optive Mega-3 PF (Active Comparator 1) | CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2)
Number analyzed (Participants) | 18 | 21 | 19 | 23
% Area of Fluorescein Darkening / sec | 0.33 [-0.55 to 1.22] | 1.71 [1.04 to 2.38] | 0.02 [-0.81 to 0.85] | 0.70 [-0.13 to 1.53]

4. Other Pre Specified Outcome: Exploratory - Subjective Symptoms - OSDI Questionnaire
Description: Change (3mo follow-up - post-run-in baseline) in Ocular Surface Disease Index (OSDI) score. The OSDI questionnaire score ranges from 0-100, with higher scores indicating more severe symptoms of Dry Eye Disease.
Time Frame: OSDI questionnaire administered once at post-run-in baseline and once at 3mo follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Systane Complete PF (Treatment) | Refresh Relieva PF (Control) | Refresh Optive Mega-3 PF (Active Comparator 1) | CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2)
Number analyzed (Participants) | 18 | 21 | 19 | 23
units on a scale | 2.88 (13.45) | 4.90 (16.31) | 2.79 (15.22) | 1.30 (9.48)

5. Other Pre Specified Outcome: Exploratory - Subjective Symptoms - SANDE
Description: Change in Symptom Assessment questionnaire iN Dry Eye (SANDE) score (3mo follow-up - post-run-in baseline)
Time Frame: SANDE questionnaire administered once at post-run-in baseline and once at 3mo follow-up visit
Population: The SANDE questionnaire was not administered to any subjects due to logistical issues.
Arm/Group | Systane Complete PF (Treatment) | Refresh Relieva PF (Control) | Refresh Optive Mega-3 PF (Active Comparator 1) | CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Other Pre Specified Outcome: Exploratory - Subjective Symptoms - DEQ-5
Description: Change in 5-Item Dry Eye Questionnaire (DEQ-5) score (3mo follow-up - post-run-in baseline)
Time Frame: DEQ-5 questionnaire administered once at post-run-in baseline and once at 3mo follow-up visit
Population: The DEQ-5 questionnaire was not administered to any subjects due to logistical issues.
Arm/Group | Systane Complete PF (Treatment) | Refresh Relieva PF (Control) | Refresh Optive Mega-3 PF (Active Comparator 1) | CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were recorded for each subject monthly for 8 months.
Arm/Group | Run-in Period Participants | Systane Complete PF (Treatment) | Refresh Relieva PF (Control) | Refresh Optive Mega-3 PF (Active Comparator 1) | CVS Health Lubricant Eye Drop (PG 0.6%) (Active Comparator 2)
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/18 | 0/21 | 0/19 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/18 | 0/21 | 0/19 | 0/23
Other Adverse Events (participants affected / at risk) | 0/81 | 0/18 | 0/21 | 0/19 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT05705518/Prot_SAP_001.pdf